CLINICAL TRIAL: NCT01329081
Title: Rehabilitation After Fast-track Total Knee Arthroplasty
Acronym: HOLEST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Kristian Larsen, Ph.D., Associate Professor, Principal Investigator, Orthopedic Research Unit, Hospital Unit West, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KL24621
Record Dates: First submitted 2010-04-27; First posted 2011-04-05 (Estimated); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Knee Arthroplasty
Keywords: Rehabilitation; Strength training; Long-term effect; Activity and participation after fast-track knee arthroplasty
MeSH Terms: conditions — Motor Activity | interventions — Rehabilitation; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Six weeks strength training in teams and patient education (Experimental)
  Interventions: Other: Postoperative rehabilitation after fast-track TKA
- Supervised home training with focus on activities (Experimental)
  Interventions: Other: Postoperative rehabilitation after fast-track TKA

INTERVENTIONS:
Other: Postoperative rehabilitation after fast-track TKA — Six weeks of strength training combined with patient education
  Other Names: Rehabilitation; Strength; Patient education
  Arms: Six weeks strength training in teams and patient education
Other: Postoperative rehabilitation after fast-track TKA — Six to eight weeks of supervised home training
  Arms: Supervised home training with focus on activities

SUMMARY:
BACKGROUND In 2008 approximately 7,700 total knee arthroplasties (TKA) were performed in Denmark. The results after TKA is in general very good, the investigators have, however, discovered that patients following fast-track TKA still have a deficit 12 months postoperatively of 5-10% in health-related quality-of-life and 15-20% in activity and participation when compared to age- and gender matched population. A postoperative rehabilitation intervention has the potential to reduce or remove this observed deficit. The current evidence of postoperative rehabilitation after TKA is, however, scares and conflicting, and no studies have shown a lasting effect beyond 3 months postoperatively.

PURPOSE The purpose of this study is to investigate if a 6-weeks postoperative rehabilitation intervention is more effective than supervised home training, and furthermore to investigate the cost-effectiveness of the intervention in a societal perspective.

MATERIALS & METHODS The study is performed as a randomized clinical trial. In total 140 patients are included in the study. Inclusion criteria are age above 18 years, patients diagnosed as having knee arthrosis, patients receiving primary elective TKA, and patients who are able to and willing transport themselves to the rehabilitation center, which demands ability to walk 50 meter, and climb 10 stair steps. Exclusion criteria are unicompartmental or revision arthroplasty, any neurological disease, knee infection, and substantial pain or functional limitation hindering rehabilitation tested by physiotherapist prior to rehabilitation start. Primary endpoint is 6 months postoperatively and primary outcome measure is change in total score by using the knee specific questionnaire Oxford Knee Score.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* patients diagnosed as having knee arthrosis
* patients receiving primary elective TKA and
* patients who are able to and willing transport themselves to the rehabilitation center, which demands ability to walk 50 meter, and climb 10 stair steps

Exclusion Criteria:

* unicompartmental or revision arthroplasty
* any neurological disease
* knee infection and
* substantial pain or functional limitation hindering rehabilitation tested by physiotherapist prior to rehabilitation start

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Oxford Knee Score | Six months postoperatively
  A disease specific questionnaire, which measures knee pain and function with 12 items. The questionnaire is sum scored with a range from 0 = worse pain and function to 48 = best pain and function

SECONDARY OUTCOMES:
EQ-5D | Twelve months postoperatively
  A generic questionnaire, which measures health-related quality-of-life (HRQOL) with 5 items. The questionnaire is scored with a range from -0.55 = worse HRQOL to 1.00 = best HRQOL

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Research Unit, Hospital Unit West, Holstebro, Denmark